CLINICAL TRIAL: NCT00251901
Title: A Randomized Double-Blind Placebo-Controlled Multi-Centre Pilot Study to Assess Symptom Response in Subjects With Pain or Discomfort in the Chest Receiving Oral Treatment With Esomeprazole 40 mg Bid for 4 Weeks.
Brief Title: Chest Pain Pilot Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9914C00001
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Chest Pain; Gastroesophageal Reflux
Keywords: Gastroesophageal reflux disease; GERD
MeSH Terms: conditions — Chest Pain; Gastroesophageal Reflux | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole

SUMMARY:
The purpose of this study is to compare the efficacy of Nexium® with placebo in relief of acid related pain or discomfort in the chest.

ELIGIBILITY:
Inclusion Criteria:

* Pain or discomfort in the chest without any identifiable cause and severe enough for the patient to seek primary medical or similar care.
* History of pain or discomfort in the chest for at least the last two weeks prior to enrollment.

Exclusion Criteria:

* Signs, symptoms or relevant investigations suggestion present symptomatic coronary heart disease.
* Patients whose pain or discomfort in the chest warrants urgent cardiac investigation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2004-05; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Relief of pain or discomfort in the chest during the last week of the 4-week treatment course.
Relief of pain or discomfort in the chest is defined as no more than one day with minimal symptoms according to the patients assessment

SECONDARY OUTCOMES:
Symptom response during the first week is based on diary cards, days 3-7.
The investigator's overall assessment of pain or discomfort in the chest during the first and fourth week.
Scores from the PRO instruments measuring pain, HRQL, anxiety and depression, health status, reflux related symptoms and overall treatment evaluation.
Adverse events, clinical laboratory variables and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Nexium Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (80):
- Canada (16):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Penticton, British Columbia
  - Research Site, Winkler, Manitoba
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Burlington, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, North York, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Charlottetown, Prince Edward Island
  - Research Site, Saint-Léonard, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Denmark (14):
  - Research Site, Charlottenlund
  - Research Site, Elsinore
  - Research Site, Esbjerg
  - Research Site, Frederiksberg
  - Research Site, Frederikssund
  - Research Site, Herning
  - Research Site, Hillerød
  - Research Site, Kolding
  - Research Site, København K
  - Research Site, København NV
  - Research Site, Odense
  - Research Site, Odense C
  - Research Site, Randers
  - Research Site, Vejle
- Germany (22):
  - Research Site, Stuttgart, Baden-Wurttemberg
  - Research Site, Augsburg, Bavaria
  - Research Site, Hanover, Lower Saxony
  - Research Site, Saarbrücken, Saarland
  - Research Site, Dresden, Saxony
  - Research Site, Halle, Saxony-Anhalt
  - Research Site, Bad Segeberg, Schleswig-Holstein
  - Research Site, Berlin, State of Berlin
  - Research Site, Augsburg
  - Research Site, Bad Segeberg
  - Research Site, Berlin
  - Research Site, Chemnitz
  - Research Site, Dillingen
  - Research Site, Dresden
  - Research Site, Görlitz
  - Research Site, Hermaringen
  - Research Site, Leipzig
  - Research Site, Löbau
  - Research Site, Magdeburg
  - Research Site, Münster
  - Research Site, Weener
  - Research Site, Wolmirstedt
- Netherlands (14):
  - Research Site, Lichtenvoorde, Gelderland
  - Research Site, Deurne, North Brabant
  - Research Site, Oldebroek, Overijssel
  - Research Site, Hoogvliet, South Holland
  - Research Site, Rijswijk, South Holland
  - Research Site, Roelofarendsveen, South Holland
  - Research Site, Rotterdam, South Holland
  - Research Site, 's-Hertogenbosch
  - Research Site, Beek en Donk
  - Research Site, Hoogwoud
  - Research Site, Huizen
  - Research Site, Nijverdal
  - Research Site, Spijkenisse
  - Research Site, Tilburg
- Norway (6):
  - Research Site, Bergen
  - Research Site, Gjøvik
  - Research Site, Hønefoss
  - Research Site, Nestun
  - Research Site, Oslo
  - Research Site, Skedsmokorset
- Sweden (8):
  - Research Site, Åkersberga
  - Research Site, Gothenburg
  - Research Site, Krokom
  - Research Site, Norrtälje
  - Research Site, Östersund
  - Research Site, Stockholm
  - Research Site, Trollhättan
  - Research Site, Umeå

REFERENCES:
- [Derived] Wade D, Cooper J, Derry F, Taylor J. Uro-Vaxom(R) versus placebo for the prevention of recurrent symptomatic urinary tract infections in participants with chronic neurogenic bladder dysfunction: a randomised controlled feasibility study. Trials. 2019 Apr 16;20(1):223. doi: 10.1186/s13063-019-3275-x. PMID 30992071
- [Derived] Flook NW, Moayyedi P, Dent J, Talley NJ, Persson T, Karlson BW, Ruth M. Acid-suppressive therapy with esomeprazole for relief of unexplained chest pain in primary care: a randomized, double-blind, placebo-controlled trial. Am J Gastroenterol. 2013 Jan;108(1):56-64. doi: 10.1038/ajg.2012.369. Epub 2012 Nov 13. PMID 23147520